CLINICAL TRIAL: NCT03184805
Title: Randomized Controlled Comparison: STOPping Versus Continuing Antiplatelet Therapy During Noncardiac Surgery and Procedures After Next Generation Drug-eluting Stent Implantation (STOP-ASP Trial)
Brief Title: STOPping Versus Continuing Antiplatelet Therapy During Noncardiac Surgery and Procedures After Next Generation Drug-eluting Stent Implantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator judged that this study can not be maintained because participant registration rate is low.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0241
Record Dates: First submitted 2017-06-07; First posted 2017-06-14 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuing aspirin (Active Comparator): Patients in the group may continue the administration of aspirin during perioperative period.
  Interventions: Drug: Continuing aspirin
- Stopping aspirin (Experimental): Patients in the group may stop medication of antiplatelet drugs during perioperative period.
  Interventions: Drug: Stopping aspirin

INTERVENTIONS:
Drug: Continuing aspirin — Subject assigned to control arm will maintain antiplatelet therapy using aspirin only at least 7 days before surgery. If subject is taking one or more antiplatelet drugs, it should be changed (for subjects taking antiplatelet drug except aspirin at enrollment) or continued (for subject taking aspirin at enrollment) with low-dose, aspirin monotherapy before surgery. Cessation of clopidogrel, ticagrelor, and prasugrel should be started at least 5 days, 3 days and 7 days before surgery, respectively. Administration of aspirin will be started at the day of cessation of previous antiplatelet regimen and maintained until third postoperative day with 100 mg once a day.
  Arms: Continuing aspirin
Drug: Stopping aspirin — Subject assigned to comparison arm will stop antiplatelet therapy before scheduled surgery or procedure. If subject is taking aspirin, clopidogrel, ticagrelor, or prasugrel, it should be discontinued for 7 days, 5 days, 3-5 days, and 7 days before surgery. Antiplatelet therapy may be restarted as previous regimen at fourth postoperative day or sooner unless significant bleeding risk or bleeding event occurs.
  Arms: Stopping aspirin

SUMMARY:
Most previous trials support the absolute increase in bleeding risk with perioperative administration of antiplatelet. Furthermore, recent studies demonstrated that perioperative major bleeding may be related to increase cardiovascular risk. The investigators will compare the efficacy and safety of continuing versus stopping antiplatelet therapy during perioperative period in patients underwent PCI(Percutaneous Coronary Intervention) with next generation DES(Drug Eluting Stent).

DETAILED DESCRIPTION:
Most current guidelines recommend to focus on continuing antiplatelet therapy (mostly with aspirin) during noncardiac surgery if possible. Although previous study showed efficacy of continuous antiplatelet therapy in reducing perioperative ischemic cardiovascular events, its effectiveness is still not clear between perioperative bleeding and ischemic risk. Most previous trials support the absolute increase in bleeding risk with perioperative administration of antiplatelet. Furthermore, recent studies demonstrated that perioperative major bleeding may be related to increase cardiovascular risk. The investigators will compare the efficacy and safety of continuing versus stopping antiplatelet therapy during perioperative period in patients underwent PCI(Percutaneous Coronary Intervention) with next generation DES(Drug Eluting Stent).

ELIGIBILITY:
Inclusion Criteria:

* Age 19-85 years
* Planning of elective noncardiac surgery or invasive procedure
* At least 1 year interval between the surgery or procedure and last PCI with next generation DES
* Currently on antiplatelet therapy

Exclusion Criteria:

* PCI with BMS(bare metal stent), 1st generation DES or bioresorbable vascular scaffold
* Total length of inserted DES in the 3 vessels >60 mm
* History of stent thrombosis
* History of coronary artery bypass grafting surgery
* Planned surgery or procedure with high bleeding risk including followings: intracranial neurosurgery, spinal canal surgery, and eye posterior chamber surgery, endoscopic mucosal resection (EMR), endoscopic submucosal dissection (ESD), ampullary resection, endoscopic retrograde cholangiopancreatography (ERCP) with endoscopic sphincterotomy plus large-balloon papillary dilation, endoscopic ultrasonography-guided fine-needle aspiration (EUS-FNA) of cystic lesions
* Left ventricular ejection fraction <40%
* Myocardial infarction within 6 months
* Any overt thromboembolism requiring medical surveillance and/or treatment
* Any clinically overt sign of hemorrhage within 3 months
* Anticoagulant therapy for any reason
* Need of continuation or discontinuation of antiplatelet therapy during surgery or procedure at the discretion of cardiologist or operator
* Any contraindication, adverse drug reaction or hypersensitivity to aspirin
* Pregnant women or women with potential childbearing
* Inability to understand or read the informed content

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
A composite of cardiac death | 1 day after discharging from the hospital
  A composite of major perioperative adverse events
nonfatal myocardial infarction (MI) | 1 day after discharging from the hospital
  A composite of major perioperative adverse events
cerebrovascular accident | 1 day after discharging from the hospital
  A composite of major perioperative adverse events
definite or probable stent thrombosis | 1 day after discharging from the hospital
  A composite of major perioperative adverse events
any revascularization and BARC(Bleeding Academic Research Consortium) ≥3 bleeding during index hospitalization for surgery or procedure | 1 day after discharging from the hospital
  A composite of major perioperative adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No